CLINICAL TRIAL: NCT00003089
Title: A Phase II Trial of Induction Paclitaxel Plus Carboplatin Followed by Thoracic Radiation Therapy With Concurrent Weekly Low-Dose Paclitaxel and Twice Weekly Amifostine for Patients With Unresectable Locally Advanced or Partially Resected Non-Small Cell Lung Cancer
Brief Title: Chemotherapy, Amifostine, and Radiation Therapy in Treating Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: TJUH-969139; CDR0000065792 (Registry Identifier: PDQ (Physician Data Query)); ALZA-97-019-ii; NCI-V97-1343
Record Dates: First submitted 1999-11-01; First posted 2004-02-19 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2006-05

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Lung Cancer
Keywords: stage II non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; adenocarcinoma of the lung; drug/agent toxicity by tissue/organ
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Amifostine; Carboplatin; Paclitaxel; Radiotherapy

INTERVENTIONS:
Drug: amifostine trihydrate
Drug: carboplatin
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Chemoprotective drugs, such as amifostine, may protect normal cells from the side effects of chemotherapy. Radiation therapy uses high-energy x-rays to damage tumor cells.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel, carboplatin, amifostine, and radiation therapy in treating patients who have unresectable locally advanced or partially resected non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxic effects and antitumor efficacy of paclitaxel plus carboplatin in patients with unresectable, intrathoracic non-small cell lung cancer (NSCLC). II. Integrate concurrent thoracic radiation therapy and weekly low dose paclitaxel into treatment of this patient population. III. Investigate a primary chemoradiotherapy treatment approach in a population of patients selected on the basis of performance status regardless of degree of weight loss. IV. Determine the effect of amifostine on the incidence of treatment nonhematologic toxic effects, specifically esophagitis, pneumonitis, and radiation dermatitis, in these patients.

OUTLINE: This is an open label study. Patients receive induction therapy comprising paclitaxel IV over 3 hours followed by carboplatin IV over 1 hour on days 1 and 21. Patients then undergo radiotherapy beginning on day 42 (or no later than day 63) daily 5 days a week for 7 weeks. Patients also receive amifostine IV over 15 minutes followed by paclitaxel IV over 3 hours weekly (day 1 each week) concurrently for the duration of radiotherapy. On 2 other days of the week, patients receive amifostine alone preceding thoracic radiotherapy. Patients are followed every 3 months for 1 year and then every 6 months until disease progression or death.

PROJECTED ACCRUAL: Approximately 15-35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven non-small cell lung cancer Adenocarcinoma Squamous cell carcinoma Large cell carcinoma Undifferentiated carcinoma Stages II-IIIB Medically inoperable stage II and IIIA Unresectable stage IIIA and IIIB Partial resection of stage IIIA or IIIB disease with histologically proven mediastinal lymph node involvement with microscopic or measurable disease Ineligible for RTOG 9410 or RTOG 9304 Men with elevated PSA no greater than 10 and no clinical evidence of prostate carcinoma are eligible No pleural effusion large enough to be visible by plain chest radiograph, unless proven to be benign Limited metastatic disease (no liver metastases) defined as: No more than 3 lung nodules outside the primary tumor suspected to be metastatic OR No more than 3 sites of suspected metastatic disease seen on bone scan or skeletal films OR 1-3 brain metastases, with plans for whole brain irradiation, with or without surgery or radiosurgery OR Single adrenal metastases not exceeding 3 cm in size

PATIENT CHARACTERISTICS: Age: Adult Performance status: ECOG 0-1 OR Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count greater than 2,000/mm3 Platelet count greater than 100,000/mm3 Hemoglobin greater than 8 g/dL Hepatic: Transaminases less than 1.5 times normal Bilirubin less than 2.0 mg/dL Renal: Creatinine less than 1.8 mg/dL Other: No concurrent severe medical problems Calorie intake of at least 1500 kcal/day No history of active malignancy within one year except: Basal cell carcinoma of the skin Squamous cell carcinoma of the skin Superficial transitional cell carcinoma of the urothelium Cervical intraepithelial neoplasia Stage I cancer of the endometrium Stage I cancer of the upper aerodigestive tract

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior thoracic radiotherapy Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-07; Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Werner-Wasik, MD, Study Chair — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania, United States